CLINICAL TRIAL: NCT05292898
Title: A Phase I, Open-label Clinical Study to Evaluate the Safety, Tolerability, and Efficacy of LCAR-AIO, a Triple-targeted Cell Preparation Targeting CD19/CD20/CD22, in Patients With Relapsed/Refractory B-cell Acute Lymphocytic Leukemia
Brief Title: A Triple-targeted Cell Preparation Targeting CD19/CD20/CD22 in Patients With Relapsed/Refractory B-cell Acute Lymphocytic Leukemia
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Achieve the proof of concept
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Collaborators: Nanjing Legend Biotech Co. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2021065
Record Dates: First submitted 2022-03-14; First posted 2022-03-23 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2024-12

CONDITIONS: Acute Lymphocytic Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LCAR-AIO Cells (Experimental): Each subject will be treated with LCAR-AIO Cells
  Interventions: Biological: LCAR-AIO Cells

INTERVENTIONS:
Biological: LCAR-AIO Cells — LCAR-AIO Cells before treatment with LCAR-AIO cells, subjects will receive a conditioning regimen (IV infusion of cyclophosphamide 300 mg/m^2 and fludarabine 30mg/m^2 once daily (QD) for 3 days.

SUMMARY:
A phase I, open-label clinical study to evaluate the safety, tolerability, and efficacy of LCAR-AIO, a triple-targeted cell preparation targeting CD19/CD20/CD22, in patients with relapsed/refractory B-cell acute lymphocytic leukemia

DETAILED DESCRIPTION:
This is an open-label, dose escalation/expansion study to assess the safety, tolerability, and efficacy of LCAR-AIO in patients ≥ 18 years of age with relapsed or refractory B-cell acute lymphocytic leukemia. Patients who meet the eligibility criteria will receive a single dose of LCAR-AIO infusion. The study will include the following sequential phases: screening, pre-treatment (cell product preparation; lymphodepleting chemotherapy), treatment and follow up.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects have fully understood the possible risks and benefits of participating in this study, are willing to follow and able to complete all trial procedures, and have signed informed consent;
2. Age 18-75 years;
3. ECOG score: 0-1;
4. Detect the expression of at least one of CD19/CD20/CD22 in leukemic cells by Flow cytometry in peripheral blood or bone marrow
5. Leukemia cells in the bone marrow >5%
6. Pathologically confirmed relapsed/refractory ALL must meet one of the following conditions:

   1. Naive patients who failed to achieve CR1 after standard chemotherapy;
   2. relapse within 12 months after CR1, or relapse after 12 months but fail to achieve CR2
   3. twice or more bone marrow relapse
   4. Philadelphia chromosomal positive (Ph+) and unable to tolerate TKI therapy, failed TKI therapy more than 2 lines, or had contraindications for TKI therapy
7. Clinical laboratory values meet screening visit criteria
8. Expected survival ≥ 3 months;

Exclusion Criteria:

1.Prior antitumor therapy with insufficient washout period; 2.CNS infiltration; Except for patients with prior CNS infiltration who are currently in remission; 3.Have received two or more targets (CD19/CD20/CD22) CAR-T cell therapy (including but not limited to sequential infusion) at any previous time, or have received CAR-T cell therapy from Camel family origin; 4.With acute or chronic graft-versus-host disease; 5.Isolated extramedullary relapse, but hepatic, spleen, or lymph node-isolated extramedullary relapse is acceptable; 6.HBsAg, HBV DNA, HCV-Ab, HCV RNA or HIV-Ab positive; 7.Pregnant or lactating women;

-

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-03-14 (Actual); Primary Completion 2025-01-10 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
Incidence, severity, and type of treatment-emergent adverse events (TEAEs) | [Time Frame: Minimum 2 years after LCAR-AIO infusion (Day 1)]
  An adverse event refers to any untoward medical occurrence in a clinical investigation subject administered a pharmaceutical product (investigational or non-investigational), which does not necessarily have a causal relationship with the treatment
Recommended Phase 2 dose (RP2D) finding | [Time Frame: 30 days after LCAR-AIO infusion (Day 1)]
  RP2D established through ATD+BOIN design
CAR positive T cells and CAR transgene levels in peripheral blood and bone marrow | [Time Frame: 2 years after LCAR-AIO infusion (Day 1)]
  CAR positive T cells and CAR transgene levels in peripheral blood and bone marrow after LCAR-AIO infusion

SECONDARY OUTCOMES:
Overall response rate (ORR) | [Time Frame: 90 days after LCAR-AIO infusion (Day 1)]
  Objective Response Rate (ORR) is defined as the proportion of subjects who achieve CR or CRi after treatment via LCAR-AIO cell infusion
Time to Response (TTR) | [Time Frame: 90 days after LCAR-AIO infusion (Day 1)]
  Time to Response (TTR) is defined as the time from the date of first infusion of LCAR-AIO to the date of the first response evaluation of the subject who has met all criteria for CR or CRi.
Duration of Response (DoR) | [Time Frame: Minimum 2 years after LCAR-AIO infusion (Day 1)]
  Duration of Remission (DoR) is defined as the time from the first documentation of remission (CR or CRi) to the first documented relapse evidence of the responders
Relapse-free survival (RFS) | [Time Frame: Minimum 2 years after LCAR-AIO infusion (Day 1)]
  Relapse-free survival (RFS) is defined as the time from the date of first infusion of the LCAR-AIO to the first documented disease relapse or death (due to any cause), whichever occurs first
Overall Survival (OS) | [Time Frame: Minimum 2 years after LCAR-AIO infusion (Day 1)]
  Overall Survival (OS) is defined as the time from the date of first infusion of LCAR-AIO to death of the subject
Incidence of anti-LCAR-AIO antibody and positive sample titer | [Time Frame: Minimum 2 years after LCAR-H93T infusion (Day 1)]
  Venous blood samples will be collected to measure LCAR-AIO positive cell concentrations and the transgenic level of LCAR-H93T, at the time points when anti-LCAR-AIO antibody serum samples are evaluated

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Beijing Gobroad BoRen Hospital, Beijing, Beijing Municipality
  - Institute of Hematology & Blood Diseases Hospital, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: No